CLINICAL TRIAL: NCT03083041
Title: A Phase II Study of SHR-1210 in Combination With Apatinib in Advanced Non-Small Cell Lung
Brief Title: A Study of SHR-1210 in Combination With Apatinib in Advanced Non-Small Cell Lung Cancer(NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-APTN-II-202-NSCLC
Record Dates: First submitted 2017-03-02; First posted 2017-03-17 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2022-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: SHR-1210; Apatinib; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR-1210，200mg,q2w plus apatinib 250mg/d (Experimental): SHR-1210 200mg, IV, Q2W and Apatinib 250mg, PO, QD
  Interventions: Biological: SHR-1210; Drug: Apatinib
- SHR-1210，200mg,q2w plus apatinib 500mg/d (Experimental): SHR-1210 200mg, IV, Q2W and Apatinib 500mg, PO, QD
  Interventions: Biological: SHR-1210; Drug: Apatinib
- SHR-1210，200mg,q2w plus apatinib 375mg/d (Experimental): SHR-1210 200mg, IV, Q2W and Apatinib 375mg, PO, QD
  Interventions: Biological: SHR-1210; Drug: Apatinib

INTERVENTIONS:
Biological: SHR-1210 — SHR-1210 will be administered as a 30-minute IV infusion Q2W at a dose of 200mg
Drug: Apatinib — Apatinib tablet will be administered orally,once daily until progression
  Other Names: Apatinib Mesylate

SUMMARY:
This is a multi-center, open-label, Phase II study of intravenous (IV) SHR-1210 at 200mg,q2w in combination with Apatinib at two dose levels in subjects with locally advanced or metastatic non-small cell lung cancer (NSCLC).

The study is composed of two parts. Part 1 of the study will determine the safety ,tolerability and pharmacokinetics of SHR-1210 in combination with Apatinib.

Part 2 includes a randomized comparison of Apatinib 250mg/d or 500mg/d plus SHR-1210 .

Subject's tumors will be screened at baseline for EGFR mutations, EML4-ALK translocation, and PD-L1 expression.But positive tumor PD-L1 expression will not be required for enrollment.

DETAILED DESCRIPTION:
SHR-1210 is a humanized monoclonal antibody against Programmed death 1(PD-1). Apatinib is a new kind of selective Vascular Endothelial Growth Factor Receptor 2(VEGFR-2) tyrosine kinase inhibitor (TKI). A disease-control rate of 61.1% and a mPFS of 4.7 months were showed in Apatinib phase II study in patients with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects >/= 18 years and </=70 years of age at the time of Informed Consent.
2. Advanced relapsed or refractory predominantly NSCLC with at least one measurable lesion according to RECIST 1.1.
3. Failure of second line of chemotherapy(Part 1);Failure of First line of chemotherapy(Part 2)
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
5. Patients must have recovered from any AEs of prior treatments before randomization.
6. Adequate bone marrow,liver and renal function as assessed by the following laboratory tests conducted within 1 week before randomization. HB ≥ 90g/L; ANC≥1.5×10E+9/L; PLT≥100×10E+9/L; ALT and AST < 1.5×ULN; TBIL ≤1×ULN; Cr ≤1.5×ULN or CL≥60 ml/min.
7. Life expectancy of at least three months.
8. Male or female participants of childbearing potential must be willing to use an adequate method of contraception starting with the first dose of study drug through 60 days for female subjects and 120 days for male subjects after the last dose of study drug.
9. Written informed consent and the willingness and ability to comply with all aspects of the protocol.

Exclusion Criteria:

1. Suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (including QT interval male ≥ 450 ms, female≥ 470 ms).
2. Severe or uncontrolled systemic disease such as clinically significant hypertension(systolic pressure >/= 140 mm Hg and/or diastolic pressure >/= 90 mm Hg), and Grade III-IV cardiac insufficiency, according to NYHA criteria or echocardiography check: LVEF<50%.
3. Factors to affect oral administration(inability to swallow tablets,GI tract resection, chronic bacillary diarrhea and intestinal obstruction).
4. Coagulation disfunction,hemorrhagic tendency or receiving anticoagulant therapy
5. >/= CTCAE 2 pneumorrhagia or >/= CTCAE 3 hemorrhage in other organs within 4 weeks.
6. Bone fracture or wounds that was not cured.
7. Arterial thrombus or phlebothrombosis within 6 months and taking anticoagulant agents.
8. Mental diseases and psychotropic substances abuse.
9. Previous treatment with an trial agent within 4 weeks
10. Proteinuria ≥ (++) or 24 hours total urine protein > 1.0 g.
11. Other coexisting malignant disease (except basal-cell carcinoma and carcinoma in situ of uterine cervix).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Part 1: Incidence and grade of adverse events (AEs) and Serious adverse events (SAEs) | up to 24 weeks
  AEs and SAEs assessed by NCI-CTCAE v4.03
Part 2:Objective response rate (ORR) per RECIST 1.1 | Up to approximately 6 months
  ORR is defined as the proportion of subjects who have achieved complete response (CR) or partial response (PR) according to RECIST 1.1

SECONDARY OUTCOMES:
Part 1: Apatinib plasma concentrations and serum SHR-1210 concentrations | Cycles 1-2(each cycle is 28 days)
  Apatinib plasma concentrations and serum SHR-1210 concentrations in Expansion cohort
Part 1:Peak Plasma Concentration (Cmax) of Apatinib and SHR-1210 | Cycles 1-2(each cycle is 28 days)
  Cmax of Apatinib and SHR-1210 in Expansion cohort
Part 1:Objective response rate (ORR) - RECIST 1.1 | Up to approximately 6 months
  ORR is defined as the proportion of subjects who have achieved complete response (CR) or partial response (PR) according to RECIST 1.1
Duration of Response (DoR) | Up to approximately 2 years
  Duration of Response (DoR) per RECIST 1.1
Progression-free survival(PFS) | Up to approximately 2 years
  PFS per RECIST 1.1
Overall survival rate at 12 months (OSR12) | Up to approximately 1 years
  OSR12 will be calculated based on Kaplan-Meier estimates of Overall survival at 12 months
Part 1: Area under the plasma concentration-time curve from time 0 to 24 hrs, AUC[0-24] | Cycles 1-2(each cycle is 28 days)
  AUC[0-24] of Apatinib and SHR-1210 in Expansion cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gao G, Ni J, Wang Y, Ren S, Liu Z, Chen G, Gu K, Zang A, Zhao J, Guo R, He J, Lin X, Pan Y, Ma Z, Wang Z, Fan M, Liu Y, Cang S, Yang X, Li W, Wang Q, Zhou C. Efficacy and safety of camrelizumab plus apatinib in previously treated patients with advanced non-small cell lung cancer harboring EGFR or ALK genetic aberration. Transl Lung Cancer Res. 2022 Jun;11(6):964-974. doi: 10.21037/tlcr-22-22. PMID 35832447